CLINICAL TRIAL: NCT01103505
Title: The HOME Study: HOme Vision Monitoring in AREDS2 for Progression to Neovascular AMD Using the ForeseeHome Device - (HOme Monitoring of the Eye)
Brief Title: HOme Vision Monitoring in AREDS2 for Progression to Neovascular AMD Using the ForeseeHome Device
Acronym: AREDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ForeseeHome AREDS2; NCT01314430 (obsolete NCT alias)
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; CNV
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ForeseeHome AMD Monitoring Device (Other): Participants in the device monitoring arm will receive a packed device at home, with instructions to install and connect the device to a modem as well as instructions for daily use of the device in addition to standard care
  Interventions: Diagnostic Test: ForeseeHome AMD Monitoring Device
- Standard care alone (control) arm (No Intervention): Standard care instruction per clinic routine for home vision monitoring to detect progression of AMD and routine eye exams

INTERVENTIONS:
Diagnostic Test: ForeseeHome AMD Monitoring Device — Earlier detection of progression from intermediate dry age-related macular degeneration to CNV between routine eye exams through home diagnostic testing with the ForeseeHome AMD Monitoring device
  Arms: ForeseeHome AMD Monitoring Device

SUMMARY:
The overall objective of this two arm randomized clinical trial (RCT) is to determine if home monitoring using the comprehensive visual field and telemedicine solution based on the ForeseeHome device in AREDS2 improves detection of progression to choroidal neovascularization (CNV) when compared with standard care.

DETAILED DESCRIPTION:
The overall objective of this two arm randomized clinical trial (RCT) is to determine if home monitoring using the comprehensive visual field and telemedicine solution based on the ForeseeHome device in AREDS2 (referred to as the ForeseeHome comprehensive solution) participants at high risk of progression to neovascular AMD improves detection of progression to choroidal neovascularization (CNV) when compared with standard care. The primary outcome of this study is presenting best corrected visual acuity (BCVA) at the time of CNV diagnosis. Secondary outcomes include time to confirmed CNV diagnosis, lesion size, lesion location (extrafoveal, juxtafoveal, or subfoveal), lesion type (occult without classic, predominantly classic or minimally classic), sensitivity and specificity, and BCVA following three consecutive months of treatment and twelve months after the initial start of CNV treatment with an intravitreal anti-VEGF agent using either ranibizumab or bevacizumab. Outcomes will be ascertained via the following specific aims:

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female participant between 55 and 90 years of age. Participants must have bilateral large drusen (at least 125 micron), or large drusen in the posterior pole in one eye (study eye) and advanced AMD (neovascular AMD or central geographic atrophy) in the fellow eye as determined by their study ophthalmologist. Likelihood, willingness, and ability to return for multiple visits (potentially within the same month) for at least 2 years.
* Participant must be English speaking and understand and sign the protocol's informed consent document.
* Participant must be able to successfully demonstrate their ability to comprehend instructions and use of the ForeseeHome device (a ForeseeHome device will be available at the clinic for the participant to demonstrate their ability).
* Participant's address to which the ForeseeHome device will be sent, if randomized to the device monitoring arm, must be located in the U.S.A.
* Study eye(s) must have best corrected visual acuity 20/60 or better (at least 54 letters).
* Ocular media sufficient to allow adequate quality fundus photography.
* Participant must be willing to have name and contact information provided to Notal Vision.
* Participant must consent to be examined by the study ophthalmologist when changes in symptoms are detected by the home-device or by standard of care or when unreliable test results occur during the usage period.
* If randomized to the device monitoring arm, participant must agree to take the device with them if staying somewhere else other than their primary residence for 14 days or more.

EXCLUSION CRITERIA:

* Participant has evidence of macular or retinal disorders other than AMD in the study eye(s).
* Participant has known adverse reaction to fluorescein dye or refuses further fluorescein angiograms.
* Participant's eye is receiving (or is expected to receive) an eye examination on a continuing basis by an eye care professional more frequently than every four months
* NonAREDS2 participant currently enrolled in another study that may likely affect adherence with The HOME Study
* Previous retinal or other ocular surgical procedures, the effects of which may now or in the future complicate assessment of the progression of AMD in the study eye.
* Chronic requirement for any systemic or ocular medication administered for other diseases
* Cataract surgery within one month of randomization.
* Participant that has any condition that would make adherence to study follow up procedures for at least one year difficult or unlikely

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1520 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Chew, MD, Study Chair — National Eye Institute (NEI)
Locations (38):
- United States (38):
  - Jones Eye Institute - UAMS, Little Rock, Arkansas
  - Shiley Eye Center - UCSD, La Jolla, California
  - Loma Linda Univ., Loma Linda, California
  - Univ. of California, Davis, Sacramento, California
  - Colorado Retina Assoc., Denver, Colorado
  - Eldorado Retina Associates, Louisville, Colorado
  - Yale Univ. Eye Center, New Haven, Connecticut
  - Univ. of Florida Health Science Center, Jacksonville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Emory Univ. Eye Center, Atlanta, Georgia
  - Georgia Retina, P.C., Decatur, Georgia
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Elman Retina Group, PA, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Ophthalmic Cons. of Boston, Boston, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Vision Research Foundation, Grand Rapids, Michigan
  - Vision Research Foundation, Royal Oak, Michigan
  - Vision Research Foundation, Traverse City, Michigan
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - Retina Research Foundation, Slingerlands, New York
  - Charlotte Eye Ear Nose and Throat Assoc, Charlotte, North Carolina
  - Duke Univ., Durham, North Carolina
  - Case Western Reserve Univ., Cleveland, Ohio
  - Retina Assoc. of Cleveland, Cleveland, Ohio
  - Pennsylvania Retina Specialists, P.C., Camp Hill, Pennsylvania
  - Penn State M.S. Hershey Med Ctr, Hershey, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Univ. of Tennessee HSC, Memphis, Tennessee
  - Texas Retina Associates, Dallas, Texas
  - Retina Consult. of Houston, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - John Moran Eye Center, Univ. of Utah, Salt Lake City, Utah
  - Univ. of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Sponsor Home Page — http://www.notalvision.com
- See also: AREDS2 page — http://www.areds2.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1970 Participants 53-90 Years of age at high risk of CNV developing were screened of these 1520 with mean age of 72.5 were enrolled at 44 clinical centers
Groups:
- Device Monitoring Arm: Participants in the device monitoring arm will receive a packed device at home, with instructions to install and connect the device to a modem as well as instructions for daily use of the device.
- Standard Care (Control) Arm: Standard care instruction per clinic routine for home vision monitoring to detect progression of AMD.
Period: Overall Study
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm
Started | 763 | 757
Completed | 739 | 737
Not Completed | 24 | 20

BASELINE CHARACTERISTICS:
Population: At baseline, all participants underwent Best corrected visual acuity testing and color fundus photography of 3 stereoscopic fields in both eyes.
Groups:
- Device Monitoring Arm: participants in the device monitoring arm will receive a packed device at home, with instructions to install and connect the device to a modem as well as instructions for daily use of the device.
  ForeseeHome
- Total: Total of all reporting groups
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm | Total
Number analyzed (Participants) | 763 | 757 | 1520
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 104 | 111 | 215
  >=65 years | 659 | 646 | 1305
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.6 (7.7) | 72.3 (7.7) | 72.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444 | 451 | 895
  Male | 319 | 306 | 625
Region of Enrollment [Number; unit: participants]
  United States | 763 | 757 | 1520

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome: Change in Visual Acuity (LogMAR Letters) From Baseline to Detection of Choroidal Neovascularization
Description: Mean change in BCVA (logMAR letters) from baseline to the time of confirmed progression to CNV in the ForeseeHome device monitoring group compared to the standard care group.
Time Frame: 2 years
Population: Patients in each study arm that progressed from intermediate AMD to CNV during the study were evaluated according to the primary and secondary endpoints. 51 of 763 patients in the device + standard care arm progressed to CNV during the trial, and 30 of 757 patients in the standard care alone arm progressed to CNV during the trial.
Measure: Mean (Standard Deviation); unit: LogMAR letters (ETDRS)
Groups:
- ForeseeHome + Standard Care at CNV Progression: Patients who progressed from intermediate AMD to CNV and who were randomized to ForeseeHome use + Standard Care at the time CNV developed
- Standard Care Alone (Control) at CNV Progression: Patients who progressed from intermediate AMD to CNV and were randomized to Standard Care alone (control arm) at the time CNV developed.
Arm/Group | ForeseeHome + Standard Care at CNV Progression | Standard Care Alone (Control) at CNV Progression
Number analyzed (Participants) | 51 | 30
LogMAR letters (ETDRS) | -7.4 (11.4) | -12.6 (16.5)

2. Secondary Outcome: Secondary Outcome: Patients Who Maintained 20/40 or Better Vision at Time of CNV Detection
Description: Percent of patients who maintained 20/40 or better vision at the time of CNV detection in each study arm
Time Frame: 2 years
Population: 51 of 763 patients progressed to CNV in the device arm and 30 of 757 patients progressed to CNV in the standard care alone arm. Patients that progressed to CNV were analyzed in this secondary analysis.
Measure: Number; unit: percentage of patients
Groups:
- Device Monitoring Arm: Participants in the ForeseeHome use + Standard Care monitoring arm who maintained 20/40 or better vision at time of CNV detection
- Standard Care (Control) Arm: Participants in the Standard Care alone monitoring arm who maintained 20/40 or better vision at time of CNV detection
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm
Number analyzed (Participants) | 51 | 30
percentage of patients | 87 | 64

3. Secondary Outcome: Secondary Outcome: Lesion Size (Total Lesion Area) at Time of Confirmed Progression to CNV
Description: Median lesion size (total lesion area) at time of confirmed progression to CNV as measured on fluorescein angiography (FA) will be compared between the two study arms. Lesion size was assessed, measured, and reported by optic disc areas, where 1 disc area = 2.54 mm^2.
Time Frame: 2 years
Population: Of 51 patients who progressed to CNV in the device arm, 39 had an FA performed, and of 30 patients who progressed to CNV in the standard care alone arm, 23 had an FA performed. Patients that progressed to CNV and had FAs performed were analyzed in this secondary analysis.
Measure: Median (Inter-Quartile Range); unit: Disc Areas
Groups:
- Device Monitoring Arm: Lesion size (total lesion area) of participants in the ForeseeHome use + Standard Care monitoring arm at time of CNV detection
- Standard Care (Control) Arm: Lesion size (total lesion area) of participants in the Standard Care alone monitoring arm at time of CNV detection
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm
Number analyzed (Participants) | 39 | 23
Disc Areas | 0.23 [0 to 0.91] | 0.70 [0 to 1.50]

4. Secondary Outcome: Secondary Outcome: Lesion Size (CNV Area) at Time of Confirmed Progression to CNV
Description: Median lesion size (CNV area) at time of confirmed progression to CNV as measured on fluorescein angiography will be compared between the two study arms. Lesion size was assessed, measured, and reported by optic disc areas, where 1 disc area = 2.54 mm^2.
Time Frame: 2 years
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Disc Areas
Groups:
- Device Monitoring Arm: Lesion size (CNV lesion area) of participants in the ForeseeHome use + Standard Care monitoring arm at time of CNV detection
- Standard Care (Control) Arm: Lesion size (CNV lesion area) of participants in the Standard Care alone monitoring arm at time of CNV detection
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm
Number analyzed (Participants) | 39 | 23
Disc Areas | 0.17 [0 to 0.69] | 0.60 [0 to 1.50]

5. Secondary Outcome: Secondary Outcome: Lesion Size (Fluid Area) at Time of Confirmed Progression to CNV
Description: Median lesion size (fluid area) at time of confirmed progression to CNV as measured on fluorescein angiography will be compared between the two study arms. Lesion size was assessed, measured, and reported by optic disc areas, where 1 disc area = 2.54 mm^2.
Time Frame: 2 years
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Disc Areas
Groups:
- Device Monitoring Arm: Lesion size (fluid area) of participants in the ForeseeHome use + Standard Care monitoring arm at time of CNV detection
- Standard Care (Control) Arm: Lesion size (fluid area) of participants in the Standard Care alone monitoring arm at time of CNV detection
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm
Number analyzed (Participants) | 51 | 30
Disc Areas | 0.55 [0 to 1.15] | 0.90 [0 to 2.20]

ADVERSE EVENTS:
Groups:
- Device Monitoring Arm: Participants in the ForeseeHome AMD device monitoring arm will receive a device for at home use, with instructions to install and connect the device to a modem as well as instructions for daily use of the device, in addition to standard care.
- Standard Care (Control) Arm: Standard care arm study participants will receive instruction per clinic routine for home vision monitoring (e.g. Amsler grid) to detect progression of AMD in addition to routine scheduled eye exams
Arm/Group | Device Monitoring Arm | Standard Care (Control) Arm
All-Cause Mortality (participants affected / at risk) | 0/763 | 0/757
Serious Adverse Events (participants affected / at risk) | 0/763 | 0/757
Other Adverse Events (participants affected / at risk) | 0/763 | 0/757

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less